CLINICAL TRIAL: NCT04434027
Title: Mother's Milk Study: Determining the Impact of Human Milk Oligosaccharides (HMOs) on Healthy Infant Growth and Development
Brief Title: The Effects of Natural Sugars in Breast Milk on Healthy Infant Growth and Development
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Children's Hospital Los Angeles (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Michael I. Goran, Principal Investigator, University of Southern California
Other Study IDs: CHLA-18-00576
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: microbiome; nutrition; obesity; growth; breastfeeding; mother; infant; cognitive development
MeSH Terms: conditions — Obesity; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Breast milk; Stool (mother and infant)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will investigate the effects of breastfeeding and breastmilk composition on infant gut microbiome development as well as obesity and cognitive outcomes. Breast milk contains certain natural sugars that can promote the growth of 'good' bacteria in the intestines and reduce the growth of harmful bacteria. The purpose of this study is to look at the effects of these natural sugars in breast milk on the infant's bacteria and the impact of this on development of obesity and cognitive outcomes by 2 years of age with plans for longer term follow up contingent upon funding.

DETAILED DESCRIPTION:
This project will examine specific factors in breast milk that may impact infant's gut microbiome development, and thereby impact their adiposity and weight gain in early life. An important early-life experience that could meaningfully impact the development of the gut microbiome, as well as future obesity risk, is breastfeeding. Breast milk has been shown to contain certain macronutrients (human milk oligosaccharides; HMOs) that not only vary greatly among women, but recent studies suggest that these factors are significant predictors of infant weight gain and adiposity. Examining early onset obesity during infancy is important because accelerated weight gain and adiposity in the first few years of life are major predictors for later obesity, and because neuronal, metabolic, and gut microbiome systems are especially vulnerable by programming from nutritional and maternal factors during this stage of life.

This study will be conducted in Los Angeles. The investigators will recruit two-hundred-and-forty mother-infant pairs. Mothers and infants will be monitored during the first 36 months of life, with sampling of breast milk (while the mother is still breast feeding) and infant and maternal stool at 1, 6, 12, 18, and 24 months of age (or as close as possible to each month). Only an infant stool sample will be collected at 36 months of age. The main outcomes of this study will be infant body weight-for-length growth during this period, as well as body composition (fat and lean mass), which will be measured by skin-fold thickness using a caliber, height, weight, and waist circumference measurements at 1, 6, 12, 18, 24, and 36 months of infant age (or as close as possible to each month). The investigators will also assess maternal and infant diet using 24-hour recalls, and maternal feeding style and infant eating behaviors using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who self-identify as Hispanic
* Mothers who have or have had singleton births
* Mothers will be recruited prior to their infant's birth or up to 1-month postpartum
* Mothers must be able/willing to understand the procedures of the study, and must be able to read English or Spanish at a 5th grade level

Exclusion Criteria:

* Physician diagnosis of a major medical illness (including type 1 or type 2 diabetes) or eating disorder in mothers
* Physical, mental, or cognitive issues that prevent participation
* Chronic use of any medication that may affect body weight or composition, insulin resistance, or lipid profiles
* Current smoking (more than 1 cigarette in the past week) or use of other recreational drugs
* Clinical diagnosis of gestational diabetes
* Pre-term/low birth weight infants, or diagnosis of any fetal abnormalities
* Mothers less than 18 years of age at the time of delivery will not be eligible as to avoid potential confounding from those subjects who might still be completing adolescent growth

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal, overweight or obese (>25 BMI kg/m2) non-diabetic Hispanic mothers (18-59yrs) and their infants (<1-36 months) from Los Angeles, CA.
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Infant weight z-scores at baseline | Baseline
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 6 months | 6 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 12 months | 12 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 18 months | 18 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 24 months | 24 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant weight z-scores at 36 months | 36 months
  Weight and length will be used to calculate weight-for-length (WLZ) and weight-for-age (WAZ) z-scores using the WHO Child Growth Standards, as recommended by the CDC for children <24 mos.
Infant skinfold thickness at baseline | Baseline
  Infant skinfold thickness will be measured in duplicate using a commercial caliper at the following sites: tricep, subscapular, suprailiac, and midthigh.
Infant skinfold thickness at 6 months | 6 months
  Infant skinfold thickness will be measured in duplicate using a commercial caliper at the following sites: tricep, subscapular, suprailiac, and midthigh.
Infant skinfold thickness at 12 months | 12 months
  Infant skinfold thickness will be measured in duplicate using a commercial caliper at the following sites: tricep, subscapular, suprailiac, and midthigh.
Infant skinfold thickness at 18 months | 18 months
  Infant skinfold thickness will be measured in duplicate using a commercial caliper at the following sites: tricep, subscapular, suprailiac, and midthigh.
Infant skinfold thickness at 24 months | 24 months
  Infant skinfold thickness will be measured in duplicate using a commercial caliper at the following sites: tricep, subscapular, suprailiac, and midthigh.
Infant skinfold thickness at 36 months | 36 months
  Infant skinfold thickness will be measured in duplicate using a commercial caliper at the following sites: tricep, subscapular, suprailiac, and midthigh.
Infant body fat measured using an EchoMRI body composition analyzer at baseline | Baseline
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 18 months | 18 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant body fat measured using an EchoMRI body composition analyzer at 24 months | 24 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant body fat in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at baseline | Baseline
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 18 months | 18 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant lean mass measured using an EchoMRI body composition analyzer at 24 months | 24 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant lean mass in grams.
Infant total body water measured using an EchoMRI body composition analyzer at baseline | Baseline
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 18 months | 18 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant total body water measured using an EchoMRI body composition analyzer at 24 months | 24 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant total body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at baseline | Baseline
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 6 months | 6 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 12 months | 12 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 18 months | 18 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.
Infant free body water measured using an EchoMRI body composition analyzer at 24 months | 24 months
  An EchoMRI infant body composition analyzer (EchoMRI LLC., Houston TX) will be used to measure infant free body water in grams.

SECONDARY OUTCOMES:
Maternal pregravid BMI | Baseline
  Maternal BMI prior to pregnancy will be derived from pregravid BMI (recall during pregnancy at baseline visit) using the equation (weight in kg)/(height in m)^2.
Maternal height at baseline | Baseline
  Height (cm) will be measured using a stadiometer.
Maternal height at 6 months | 6 months
  Height (cm) will be measured using a stadiometer.
Maternal height at 12 months | 12 months
  Height (cm) will be measured using a stadiometer.
Maternal height at 18 months | 18 months
  Height (cm) will be measured using a stadiometer.
Maternal height at 24 months | 24 months
  Height (cm) will be measured using a stadiometer.
Maternal weight at baseline | Baseline
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 6 months | 6 months
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 12 months | 12 months
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 18 months | 18 months
  Weight (kg) will be measured using a portable digital scale.
Maternal weight at 24 months | 24 months
  Weight (kg) will be measured using a portable digital scale.
Maternal BMI at baseline | Baseline
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 6 months | 6 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 12 months | 12 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 18 months | 18 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Maternal BMI at 24 months | 24 months
  Body Mass Index (BMI) will be calculated based on the equation (weight in kg)/(height in m)^2.
Infant length at baseline | Baseline
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 6 months | 6 months
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 12 months | 12 months
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 18 months | 18 months
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 24 months | 24 months
  Infant length (cm) will be measured using an infant measure mat.
Infant length at 36 months | 36 months
  Infant length (cm) will be measured using an infant measure mat.
Infant weight at baseline | Baseline
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 6 months | 6 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 12 months | 12 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 18 months | 18 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 24 months | 24 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Infant weight at 36 months | 36 months
  Infant weight (kg) will measured using a portable digital scale. For infants that need to be held, weight will be calculated as follows: (combined mother + infant weight) - (mother only weight).
Maternal systolic and diastolic blood pressure at baseline | Baseline
  Sitting systolic and diastolic blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal systolic and diastolic blood pressure at 6 months | 6 months
  Sitting systolic and diastolic blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal systolic and diastolic blood pressure at 12 months | 12 months
  Sitting systolic and diastolic blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal systolic and diastolic blood pressure at 18 months | 18 months
  Sitting systolic and diastolic blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal systolic and diastolic blood pressure at 24 months | 24 months
  Sitting systolic and diastolic blood pressure will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at baseline | Baseline
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 6 months | 6 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 12 months | 12 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 18 months | 18 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal resting heart rate at 24 months | 24 months
  Sitting heart rate will be measured on the right arm after the subject has rested quietly for 5 minutes using a digital blood pressure monitor (Omron 3-series).
Maternal diet at baseline | Baseline
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Maternal diet at 6 months | 6 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Maternal diet at 12 months | 12 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Maternal diet at 18 months | 18 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Maternal diet at 24 months | 24 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at baseline | Baseline
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at 6 months | 6 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at 12 months | 12 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at 18 months | 18 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at 24 months | 24 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Infant diet at 36 months | 36 months
  24-hour diet recalls will be conducted for one week day and one weekend day. Mothers will be interviewed to report on their infant's food intake. Dietary intake will be collected and analyzed using the most current version of the Nutrition Data System for Research software (NDSR) which has been used extensively in Hispanic studies.
Maternal beverage recall during last trimester of pregnancy | Baseline
  Beverage intake of sugar-sweetened beverages and water will be recalled for a typical week during the last trimester of pregnancy. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day.
Maternal beverage recall at baseline | Baseline
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day.
Maternal beverage recall at 6 months | 6 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day.
Maternal beverage recall at 12 months | 12 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day.
Maternal beverage recall at 18 months | 18 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day.
Maternal beverage recall at 24 months | 24 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day.
Infant beverage recall at baseline | Baseline
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day. Mothers will be interviewed to report on their infant's beverage intake.
Infant beverage recall at 6 months | 6 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day. Mothers will be interviewed to report on their infant's beverage intake.
Infant beverage recall at 12 months | 12 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day. Mothers will be interviewed to report on their infant's beverage intake.
Infant beverage recall at 18 months | 18 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day. Mothers will be interviewed to report on their infant's beverage intake.
Infant beverage recall at 24 months | 24 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day. Mothers will be interviewed to report on their infant's beverage intake.
Infant beverage recall at 36 months | 36 months
  Beverage intake of sugar-sweetened beverages and water will be recalled for 1 week. Beverage recalls will indicate how many days each beverage was consumed, and how much was consumed each day. Mothers will be interviewed to report on their infant's beverage intake.
Infant feeding score assessed by Infant Feeding Questionnaire at baseline | Baseline
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 6 months | 6 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 12 months | 12 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 18 months | 18 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding score assessed by Infant Feeding Questionnaire at 24 months | 24 months
  Infant feeding score will be assessed using the Baughcum Infant Feeding Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: concern about the child undereating or becoming underweight; concern about infant's hunger; awareness of infant's cues; concern about the infant becoming overweight or overeating; feeding the infant on schedule; using food to calm the infant; social interaction during feeding.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at baseline | Baseline
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 6 months | 6 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 12 months | 12 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 18 months | 18 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant feeding style score assessed by Infant Feeding Style Questionnaire at 24 months | 24 months
  Infant feeding style score will be assessed using the Thompson Infant Feeding Style Questionnaire. Questions are scored using the following scale: 1-5; disagree, slightly disagree, neutral, slightly agree, agree. Average scores will be used to determine the following constructs: laissez-faire; pressuring; restrictive; responsive; and indulgent.
Infant behavior score assessed by Infant Behavior Questionnaire at baseline | Baseline
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant behavior score assessed by Infant Behavior Questionnaire at 6 months | 6 months
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant behavior score assessed by Infant Behavior Questionnaire at 12 months | 12 months
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant behavior score assessed by Infant Behavior Questionnaire at 18 months | 18 months
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant behavior score assessed by Infant Behavior Questionnaire at 24 months | 24 months
  Infant behavior score will be assessed using the Rothbart Infant Behavior Questionnaire. Questions are scored using the following scale: 1-7; never, very rarely, less than half the time, about half the time, more than half the time, almost always, always. Composite scores will be used to determine the following constructs: surgency/extroversion; negative affectivity; and orienting/regulation.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at baseline | Baseline
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at 6 months | 6 months
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at 12 months | 12 months
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at 18 months | 18 months
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant eating behavior score assessed by Baby Eating Behavior Questionnaire at 24 months | 24 months
  Infant eating behavior score will be assessed using the Llewellyn Baby Eating Behavior Questionnaire. Questions are scored using the following scale: 1-5; never, rarely, sometimes, often, always. Average scores will be used to determine the following constructs: food responsiveness; satiety responsiveness; slowness in eating; enjoyment of food; and general appetite.
Infant diet score assessed by Infant Diet Questionnaire at baseline | Baseline
  Infant diet will be assessed using a questionnaire which inquires about breastfeeding frequency and duration, formula type/brand/frequency, and consumption of fruit, vegetables, meat, fried foods, juice, and sweetened drinks.
Infant diet score assessed by Infant Diet Questionnaire at 6 months | 6 months
  Infant diet will be assessed using a questionnaire which inquires about breastfeeding frequency and duration, formula type/brand/frequency, and consumption of fruit, vegetables, meat, fried foods, juice, and sweetened drinks.
Infant diet score assessed by Infant Diet Questionnaire at 12 months | 12 months
  Infant diet will be assessed using a questionnaire which inquires about breastfeeding frequency and duration, formula type/brand/frequency, and consumption of fruit, vegetables, meat, fried foods, juice, and sweetened drinks.
Infant diet score assessed by Infant Diet Questionnaire at 18 months | 18 months
  Infant diet will be assessed using a questionnaire which inquires about breastfeeding frequency and duration, formula type/brand/frequency, and consumption of fruit, vegetables, meat, fried foods, juice, and sweetened drinks.
Infant diet score assessed by Infant Diet Questionnaire at 24 months | 24 months
  Infant diet will be assessed using a questionnaire which inquires about breastfeeding frequency and duration, formula type/brand/frequency, and consumption of fruit, vegetables, meat, fried foods, juice, and sweetened drinks.
Infant development assessed by the Bayley Scales of Infant and Toddler Development at 24 months | 24 months
  Infant development will be assessed using the Bayley Scales of Infant and Toddler Development - Third Edition (BSID-3). This test is designed to assess cognitive, language, motor, social-emotional, and adaptive behavior development in infants and toddlers. This test will be administered and interpreted by trained research personnel. Subscale scores each range from 1 - 19, with higher scores indicating higher performance. Scores from 8 to 12 are considered average.
Infant Magnetic Resonance Imaging (MRI) brain scan at baseline | Baseline
  Infant brain will be scanned using Magnetic Resonance Imaging (MRI) to measure structure and function.
Infant Magnetic Resonance Imaging (MRI) brain scan at 6 months | 6 months
  Infant brain will be scanned using Magnetic Resonance Imaging (MRI) to measure structure and function.
Infant development assessed by the Adaptive Behavior Assessment System at 36 months | 36 months
  Infant emotional and adaptive development will be assessed using the Adaptive Behavior Assessment System (ABAS).
Breast milk composition at baseline | Baseline
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 6 months | 6 months
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 12 months | 12 months
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 18 months | 18 months
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Breast milk composition at 24 months | 24 months
  Breast milk will be collected from mothers at least 1½ hours since the last feeding and while the mother has fasted at least 1 hour. Samples will be analyzed for glucose, fructose, galactose, lactose and sucrose by mass spectrometry. Samples will be available for analysis of insulin, leptin, and energy content.
Infant gut microbiome at baseline | Baseline
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Infant gut microbiome at 6 months | 6 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Infant gut microbiome at 12 months | 12 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Infant gut microbiome at 18 months | 18 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Infant gut microbiome at 24 months | 24 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Infant gut microbiome at 36 months | 36 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Maternal gut microbiome at baseline | Baseline
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Maternal gut microbiome at 6 months | 6 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Maternal gut microbiome at 12 months | 12 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Maternal gut microbiome at 18 months | 18 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.
Maternal gut microbiome at 24 months | 24 months
  Stool samples will be collected in OmniGUT gene kits and aliquoted to be stored at -80oC. Gut microbes will be analyzed using 16S sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, PhD, Principal Investigator — University of Southern California; Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States